CLINICAL TRIAL: NCT04224649
Title: A Single Center, Randomized, Subject & Evaluator-blind, Matched Pairs, Active-controlled Design Pivotal Study to Evaluate the Efficacy and Safety of Injection With HARA as Compared to Restylane® Lidocaine in Temporary Correction of Nasolabial Folds
Brief Title: To Evaluate the Efficacy and Safety of Injection With HARA as Compared to Restylane® Lidocaine in Temporary Correction of Nasolabial Folds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huons Co., Ltd. (Industry)
Collaborators: Humedix Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-055
Record Dates: First submitted 2019-09-05; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Nasolabial FOLD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Device Group(HARA filler) (Experimental)
  Interventions: Device: HARA Filler(Hyaluronic acid Filler)
- Comparator Group(Restylane® Lidocaine) (Active Comparator)
  Interventions: Device: Restylane® Lidocaine

INTERVENTIONS:
Device: HARA Filler(Hyaluronic acid Filler) — The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Arms: Test Device Group(HARA filler)
Device: Restylane® Lidocaine — The same participants received the experimental device and the active comparator device at the same time (left and right sides of face).
  Arms: Comparator Group(Restylane® Lidocaine)

SUMMARY:
* Investigational Device : HARA (Hyaluronic Acid Filler)
* Title : A Single center, Randomized, Subject & Evaluator-blind, Matched pairs, Active-controlled design Pivotal study to Evaluate the Efficacy and Safety of Injection with HARA as Compared to Restylane® Lidocaine in temporary Correction of Nasolabial folds
* Sites and investigators : Chung-ang University Hospital(Seoul), Beom-Joon Kim, M.D, Ph.D
* Objective : To compare the non-inferiority of HARA with Restylane® Lidocaine for evaluation of the efficacy and safety on Nasolabial Folds

ELIGIBILITY:
Inclusion Criteria:

1. Those who agreed to this treatment and signed the Informed Consent Form
2. Those who are 19 years old or more and desire to take correction of nasolabial folds
3. Those who have an intention of refraining from other cosmetic treatment(other filler injection, laser or chemical peeling, Botox injection or wrinkle reduction) during the clinical study period
4. Those whose Wrinkle Severity Rating Scale (WSRS) is more than 2 points at least

Exclusion Criteria:

1. Those who are sensitive to lidocaine or other amide anesthesia
2. Those who are sensitive to control device
3. Those who are pregnant or lactating, or expect pregnancy
4. Those who are judged by the subinvestigator to be improper for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Assessment By independent evaluator | Week 24 From baseline Visit(=Investigational Device Injection)
  Wrinkle Severity Rating Scale (WSRS, Wrinkle severity Rating scale)
  * Grade 1: Absent, Grade 2: Mild, Grade 3: Moderate, Grade 4: Severe, Grade 5: Extereme

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided